CLINICAL TRIAL: NCT03177733
Title: Evaluation of a Breast Double Block Analgesia for the Mastectomy With Radical Axillary Lymphadenectomy Surgery
Status: Completed | Type: Observational
Sponsor: Maison de Santé Prostestante de Bordeaux Bagatelle (Other)
Responsible Party: Principal Investigator, Dr Claude-Charles Balick-Weber, Principal Investigator, Maison de Santé Prostestante de Bordeaux Bagatelle
Other Study IDs: Evaluation of breast biblock 2
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Mastectomy
Keywords: breast surgery; acute pain; regional anesthesia
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Evaluation of a breast double block — we made an association of the serratus block and the PIF block, which allows for a complete block of both the laterals branches of intercostal nerves (with the serratus block) and of anterior branches of intercostal nerves (with the PIF block). Therefore, this association of blocks may lead to a complete analgesia of the breast, while the serratus block alone only allows for an analgesia of the lateral part of the breast.
  The objective is to analyze this technique through a collection form that evaluates the satisfaction and post-operative morphine consumption of women receiving this association before a general anesthesia for a unilateral mastectomy with homolateral total lymphadenectomy.
  This is a purely observational study that assesses our current practice in this type of surgery.

SUMMARY:
This study evaluates the efficacy of the the pecto-intercostal fascial plane block (PIF block) for the anesthesia of the intercostal nerves anterior branches and assesses the association of the serratus block with a PIF block for the breast surgery.

To obtain a correct prospective clinical trial completion we have to begin a new series of inclusion.

DETAILED DESCRIPTION:
Breast surgery is one of the most painful post-operative surgery. This surgery is well known to induce postoperative chronic pain. The paravertebral block, because of its efficacy and less invasive nature than epidural analgesia, is quickly becoming the reference technique for pain management of major breast surgery.

Peripheral regional anesthesia for the breast surgery appeared in the past few years. Among these techniques are the PEC block, Serratus block and more recently the pecto-intercostal fascial plane block (PIF block).

Currently in our hospital in every day's practice, we made an association of the serratus block and the PIF block, which allows for a complete block of both the laterals branches of intercostal nerves (with the serratus block) and of anterior branches of intercostal nerves (with the PIF block). Therefore, this association of blocks may lead to a complete analgesia of the breast, while the serratus block alone only allows for an analgesia of the lateral part of the breast.

This technique was described by Fajardo et al. They evoked the possibility of the association serratus and PIF blocks and described this technique with a patient, but to our knowledge no evaluation of the efficacy of this procedure was made.

The objective of your study is to analyze this technique through a collection form that evaluates the satisfaction and post-operative morphine consumption of women receiving this association of blocks before a general anesthesia for a unilateral mastectomy with homolateral total lymphadenectomy.

This is a purely observational study that assesses our current practice in this type of surgery.

we already included a patient series but the clinical trial registration was made to late to do it correctly. To obtain a correct prospective clinicaltrials registration completion we have to begin a new series of inclusion.

ELIGIBILITY:
Inclusion Criteria:

* total mastectomy surgery with a complete axillary lymph nodes removal

Exclusion Criteria:

* age under 18
* contraindication to the surgery
* refusal of the protocol by the patient

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All patients included in the study have had a total mastectomy surgery with a complete axillary lymph nodes removal.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
postoperative morphine consumption until 72 hours after the surgery. | 3 days
  The primary goal of the study is to evaluate the postoperative morphine consumption until 72 hours after the surgery.

SECONDARY OUTCOMES:
Pain levels during the first 72 hours. | 3 days
  Pain levels on a numeric pain rating scale were recorded at rest and with arm mobilization during the first 72 hours.
Level of comfort during the first 72 hours | 3 days
  level of comfort during the first 72 hours was recorded (the 4 levels-scale used was: excellent, good, medium and bad).

CONTACTS AND LOCATIONS:
Overall Officials: Claude-charles Balick-weber, Principal Investigator — Maison de Santé Protestante de Bordeaux-Bagatelle
Locations (1):
- Maison de Santé Protestante de Bordeaux-Bagatelle, Talence, Aquitaine, France

IPD SHARING:
Plan to Share IPD: Undecided